CLINICAL TRIAL: NCT00170560
Title: Impact of Gender on Infected Hospitalized Patients
Brief Title: Impact of Gender on Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 01-337
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2007-10

CONDITIONS: Hospital-acquired Infections
Keywords: hospital, acquired, infections, mortality
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to better understand the relationship between gender (being a man or a woman), infections caught in the hospital, and serious illness. Five hundred seventy patients 18 years of age or older who are critically (seriously) ill and admitted to the Intensive Care Unit (ICU) for at least 48 hours will participate in this study. Patients will be studied while receiving regular ICU treatment according to local standards. Blood specimens will come from patients either as wasted blood (University of Virginia) or blood collected from patients specifically for the study (Vanderbilt University). All patients will be followed daily until death or discharge from the ICU. The researchers believe that they will find a similar risk of infection for men and women overall.

DETAILED DESCRIPTION:
The purpose of this study is to gain knowledge that will be used to design further interventional studies to better define beneficial therapies related to gender, infection, and critical illness, such as modulation of hormone levels in a sex-specific manner. This is a two-year observational study in which approximately a total of 570 patients will be enrolled. All patients will be 18 years of age or older and admitted to the Intensive Care Unit (ICU) for at least 48 hours. Patients will be studied while receiving accepted and approved therapy according to local standards. Data obtained will be that which would normally be considered part of a standard complete medical history. Specimens will come from patients either as wasted blood (University of Virginia) or blood drawn from patients specifically for this purpose (Vanderbilt University). The maximum blood removed will be 30 ml twice weekly and is considered a minor risk. All specimens analyzed, regardless of institution, are done so in a blinded manner, identified only by study number and specimen number or through password and encryption protected servers when communicated electronically. Since the cohort is comprised of all patients admitted to an ICU, recruitment in the normal sense is not practical. An initial comparison of demographic data, severity of illness, frequency of comorbidities, hormone and cytokine levels, and outcome variables will be compared between males and females treated for infection. All patients will be followed daily until death or discharge from the ICU. It is anticipated that a similar risk of infection for men and women overall will be determined. Specific Aim I of the study is to prospectively determine and compare the incidence of and associated mortality from hospital-acquired infections in a large, critically-ill population of pre-menopausal women, post-menopausal women, and men after controlling for multiple pre-defined confounding variables. The Specific Aim II of the study is to determine the relationship between sex hormonal status, systemic cytokine levels, and the incidence of and outcome from hospital-acquired infections, as well as the relative contribution of infection and end-of-life decisions to outcome in subjects dying under study.

ELIGIBILITY:
Inclusion Criteria:

1. All patients >= 18 years old admitted to the ICU for >= 48 hours.

Exclusion Criteria:

1. Age < 18 years old.
2. Death or discharge within 48 hours of ICU admission.
3. Patients not on a surgical service.
4. Patients admitted with a primary diagnosis of burns.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Guidry CA, Swenson BR, Davies SW, Dossett LA, Popovsky KA, Bonatti H, Evans HL, Metzger R, Hedrick TL, Tache-Leon CA, Hranjec T, Chaudry IH, Pruett TL, May AK, Sawyer RG. Sex- and diagnosis-dependent differences in mortality and admission cytokine levels among patients admitted for intensive care. Crit Care Med. 2014 May;42(5):1110-20. doi: 10.1097/CCM.0000000000000139. PMID 24365862
- [Derived] Heffernan DS, Dossett LA, Lightfoot MA, Fremont RD, Ware LB, Sawyer RG, May AK. Gender and acute respiratory distress syndrome in critically injured adults: a prospective study. J Trauma. 2011 Oct;71(4):878-83; discussion 883-5. doi: 10.1097/TA.0b013e31822c0d31. PMID 21986736
- [Derived] Kauffmann RM, Norris PR, Jenkins JM, Dupont WD, Torres RE, Blume JD, Dossett LA, Hranjec T, Sawyer RG, May AK. Trends in estradiol during critical illness are associated with mortality independent of admission estradiol. J Am Coll Surg. 2011 Apr;212(4):703-12; discussion 712-3. doi: 10.1016/j.jamcollsurg.2010.12.017. PMID 21463817
- [Derived] Hranjec T, Swenson BR, Dossett LA, Metzger R, Flohr TR, Popovsky KA, Bonatti HJ, May AK, Sawyer RG. Diagnosis-dependent relationships between cytokine levels and survival in patients admitted for surgical critical care. J Am Coll Surg. 2010 May;210(5):833-44, 845-6. doi: 10.1016/j.jamcollsurg.2009.12.042. PMID 20421061
- [Derived] Collier B, Dossett L, Shipman J, Day M, Lawson G, Sawyer R, May A. Visceral adiposity is not associated with inflammatory markers in trauma patients. J Trauma. 2010 Jan;68(1):57-61. doi: 10.1097/TA.0b013e3181c40262. PMID 20065758
- [Derived] Dossett LA, Redhage LA, Sawyer RG, May AK. Revisiting the validity of APACHE II in the trauma ICU: improved risk stratification in critically injured adults. Injury. 2009 Sep;40(9):993-8. doi: 10.1016/j.injury.2009.03.004. Epub 2009 Jun 16. PMID 19535054
- [Derived] Dossett LA, Dageforde LA, Swenson BR, Metzger R, Bonatti H, Sawyer RG, May AK. Obesity and site-specific nosocomial infection risk in the intensive care unit. Surg Infect (Larchmt). 2009 Apr;10(2):137-42. doi: 10.1089/sur.2008.028. PMID 19388836
- [Derived] Dossett LA, Swenson BR, Evans HL, Bonatti H, Sawyer RG, May AK. Serum estradiol concentration as a predictor of death in critically ill and injured adults. Surg Infect (Larchmt). 2008 Feb;9(1):41-8. doi: 10.1089/sur.2007.037. PMID 18363467
- [Derived] Dossett LA, Swenson BR, Heffernan D, Bonatti H, Metzger R, Sawyer RG, May AK. High levels of endogenous estrogens are associated with death in the critically injured adult. J Trauma. 2008 Mar;64(3):580-5. doi: 10.1097/TA.0b013e31816543dd. PMID 18332796
- [Derived] May AK, Dossett LA, Norris PR, Hansen EN, Dorsett RC, Popovsky KA, Sawyer RG. Estradiol is associated with mortality in critically ill trauma and surgical patients. Crit Care Med. 2008 Jan;36(1):62-8. doi: 10.1097/01.CCM.0000292015.16171.6D. PMID 18090358